CLINICAL TRIAL: NCT00002539
Title: A RANDOMISED TRIAL OF CHEMOTHERAPY WITH OR WITHOUT GRANULOCYTE COLONY-STIMULATING FACTOR IN OPERABLE OSTEOSARCOMA
Brief Title: Combination Chemotherapy and Surgery With or Without G-CSF in Treating Patients With Osteosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-80931; EOI-80931; EORTC-80931; MRC-BO06; EU-93024
Record Dates: First submitted 1999-11-01; First posted 2003-04-10 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma
Keywords: localized osteosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Filgrastim; Cisplatin; Doxorubicin

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as G-CSF may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. It is not yet known whether chemotherapy and surgery plus G-CSF is more effective than chemotherapy and surgery alone in treating patients with osteosarcoma.

PURPOSE: Randomized phase III trial to compare the effectiveness combination chemotherapy and surgery with or without G-CSF in treating patients who have newly diagnosed osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall and disease-free survival of patients with newly diagnosed osteosarcoma of the extremity treated with conventional vs intensive cisplatin and doxorubicin with or without filgrastim (G-CSF) before and after definitive surgery.
* Compare the toxicity of these regimens in these patients.
* Compare the response in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive conventional doxorubicin (DOX) IV over 4 hours on days 1-3 and cisplatin (CDDP) IV continuously on day 1. Treatment continues every 3 weeks for 2 courses. At week 6, patients undergo amputation or local resection based on pretherapy imaging and response to chemotherapy. Beginning 2 weeks after surgery, patients receive 4 additional courses of conventional chemotherapy.
* Arm II: Patients receive intensive DOX and CDDP as above on day 1 plus filgrastim (G-CSF) subcutaneously on days 4-13. Treatment continues every 2 weeks for 3 courses. At week 6, patients undergo definitive surgery as in arm I. Beginning 2 weeks after surgery, patients receive 3 additional courses of intensive DOX and CDDP with G-CSF.

Patients who experience disease progression during preoperative chemotherapy undergo surgery earlier than scheduled and complete all scheduled chemotherapy (6 courses) after surgery, at the discretion of the surgeon and oncologist. Within 4 weeks after limb-sparing procedure, patients with inadequate margins undergo amputation, followed 2 weeks later by chemotherapy.

Patients are followed monthly for 6 months, every 2 months for 6 months, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven resectable osteosarcoma of the long bone of an extremity
* No parosteal (juxtacortical), periosteal, Pagetoid, or post-irradiation sarcoma
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 40 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3 OR
* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.2 mg/dL

Renal:

* Glomerular filtration rate at least 60 mL/min

Cardiovascular:

* No history of cardiac dysfunction

Other:

* No other prior or concurrent malignancy except basal cell skin cancer OR
* Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No prior therapy

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 1993-08; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne A. Nooij, MD, Study Chair — Leiden University Medical Center; Ian J. Lewis, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (16):
- Belgium (4):
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
- Centre Eugene Marquis, Rennes, France
- Netherlands (5):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Emma Kinderziekenhuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil-Centro de Lisboa, Lisbon, Portugal
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- St. James's Hospital, Leeds, England, United Kingdom

REFERENCES:
- [Result] Lewis IJ, Nooij MA, Whelan J, Sydes MR, Grimer R, Hogendoorn PC, Memon MA, Weeden S, Uscinska BM, van Glabbeke M, Kirkpatrick A, Hauben EI, Craft AW, Taminiau AH; MRC BO06 and EORTC 80931 collaborators; European Osteosarcoma Intergroup. Improvement in histologic response but not survival in osteosarcoma patients treated with intensified chemotherapy: a randomized phase III trial of the European Osteosarcoma Intergroup. J Natl Cancer Inst. 2007 Jan 17;99(2):112-28. doi: 10.1093/jnci/djk015. PMID 17227995
- [Result] Lewis IJ, Nooij M: Chemotherapy at standard or increased dose intensity in patients with operable osteosarcoma of the extremity: a randomised controlled trial conducted by the European Osteo Sarcoma Intergroup (ISRCTN 86294690). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3281, 816, 2003.